CLINICAL TRIAL: NCT02418065
Title: Multimodal Therapeutic Approach by Exercise, Oral Nutritional Supplementation, Omega 3 and Androgen in Undernourished Maintenance Hemodialysis Patients (AMERICANO)
Brief Title: Multimodal Therapeutic Approach in Undernourished Maintenance Hemodialysis Patients (AMERICANO)
Acronym: AMERICANO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Human Nutrition Research Center Rhône-Alpes (Unknown); Société Francophone Nutrition Clinique et Métabolisme (Other); Nutricia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHU-0231
Record Dates: First submitted 2015-04-03; First posted 2015-04-16 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Kidney Failure
Keywords: Physical exercises; Oral nutritional supplementation; Multimodal; Hemodialysis; Protein-Energy Wasting
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity | interventions — Testosterone; Dietary Supplements; Fatty Acids, Omega-3

ARMS (2):
- treated group (Experimental): testosteron, oral nutritional supplementation, n3 polyunsaturated fatty acid, training on ergonomic bicycle
  Interventions: Other: training on ergonomic bicycle; Drug: Testosterone; Drug: Oral nutritional supplementation; Drug: n3 polyunsaturated fatty acid
- control group (Other): oral nutritional supplementation
  Interventions: Drug: Oral nutritional supplementation

INTERVENTIONS:
Other: training on ergonomic bicycle
  Arms: treated group
Drug: Testosterone
  Arms: treated group
Drug: Oral nutritional supplementation
Drug: n3 polyunsaturated fatty acid
  Arms: treated group

SUMMARY:
The aim of the study is to evaluate a 3 months integrated multimodal therapeutic approach including exercise training program with ergocycle during dialysis sessions, oral nutritional supplementation, omega 3 and androgen, on effort tolerance and quality of life of under-nourish maintenance hemodialysis Chronic Kidney Disease (CKD) patient.

DETAILED DESCRIPTION:
The aim of the study is to evaluate a 3 months integrated multimodal therapeutic approach including exercise training program with ergocycle during dialysis sessions, oral nutritional supplementation, omega 3 and androgen, on effort tolerance and quality of life of under-nourish maintenance hemodialysis Chronic Kidney Disease (CKD) patient.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patient since at least 6 month
* Patient aged 18 years or older
* Written consent to participate in the study
* No acute infection or hospitalization
* Opinion of Cardiologist saying there is no known evidence against the evaluation of the maximum exercise capacity
* Protein-energy wasting diagnosed if at least two of this characteristics are present
* Serum albumin <3.8 g per 100 ml (Bromcresol Green)
* Serum prealbumin (transthyretin) <30mg per 100 ml
* Reduce body mass (BMI <23)
* Unintentional 10% weight loss over 6 months
* Lean body mass index < 10th percentile

Exclusion Criteria:

* Presence of comorbidity which compromising the survival within 6 month
* Unintentional low DEI <20 kcal kg_1 day_1
* HIV or HCV positive
* History of hormone dependent cancer
* Suspected or confirmed prostate cancer or breast carcinoma
* Known hypersensitivity for testosterone
* Presence or history of hepatic tumor
* Inability to follow the rehabilitation program
* Inadequate dialysis dosage (<12 hours / week or Kt/V index< 1,2) Pregnant or planning pregnancy and lactating women during study period
* Adult patient protected by law
* Patient who don't sign his informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Change of physical endurance on bicycle | At months 3 and 15 after inclusion
  Physical endurance on bicycle at intermediate power between maximal power and ventilatory threshold power (Pmax+Pthreshold)/2

SECONDARY OUTCOMES:
Transthyrin serum concentration evolution | at day 1
  (Unit of Measure: g/L)
Health-related quality of life assessment using SF-36 scale and KDQOL | at day 1
Karnofsky score | at ady 1
Maximal power on bicycle | at day 1
  Unit of Measure: Watt
Nutritional parameters | at day 1
  weight (Kg)
serum levels of albumin (g/L) | at day 1
determination of urea (mmol/L) | at day 1
determination of creatinine(µmol/L) | at 1 year
Body composition | at day 1
  (evaluated by bioimpedance)

CONTACTS AND LOCATIONS:
Overall Officials: Noël CANO, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133